CLINICAL TRIAL: NCT04984252
Title: Testing a Brief and Low Intensity Self-compassion Intervention for State Body Shame Among Adult Women: a Randomized Controlled Trial
Brief Title: Testing a Brief and Low Intensity Self-compassion Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Fidan Turk, Principal investigator, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 040360
Record Dates: First submitted 2021-07-08; First posted 2021-07-30 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Body Image Disturbance; Body Image; Shame
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Only Active components (Active Comparator): 15 minutes, once
  Interventions: Behavioral: Self-compassion comprising compassionate body scan-1, compassion body scan-2 and short noticing practice
- Inactive components (Sham Comparator): 15 minutes, once
  Interventions: Behavioral: Self-compassion comprising self-compassion break, loving kindness meditation, and breathing exercise.
- Distraction group (Placebo Comparator): 15 minutes, once
  Interventions: Behavioral: Distraction group

INTERVENTIONS:
Behavioral: Self-compassion comprising compassionate body scan-1, compassion body scan-2 and short noticing practice — This intervention includes 3 short meditations that are identified as the active component in the previous study (ID: NCT04665167)
  Arms: Only Active components
Behavioral: Self-compassion comprising self-compassion break, loving kindness meditation, and breathing exercise. — This intervention includes 3 short meditations that are identified as the inactive component in the previous study (ID: NCT04665167)
  Arms: Inactive components
Behavioral: Distraction group — Participants will be asked to listen recording on irrelevant topic.
  Arms: Distraction group

SUMMARY:
The investigators' recent feasibility trial of a self-compassion and active control intervention showed that the self-compassion intervention was promising in reducing state body shame during a 40-minute intervention session. There were three time points where the reduction in the body shame level was significant, indicating three active components in the intervention that led to significant reduction in state body shame. It is unclear if a shorter self-compassion intervention based on only the active components would be as effective as the longer intervention at reducing state body shame. Such a short intervention then could be used as an in-session change method (15-20 mins) as part of a larger package, or as a homework exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Self-identified women
* Be able to use a computer and have an Internet connection

Exclusion Criteria:

* Insufficient knowledge of English
* Learning disability or psychiatric illness requiring secondary care intervention
* Male
* Under 18 years old
* No access to a tablet or computer with an internet connection
* Body mass index below 18.5

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified women
Enrollment: 69 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline Subjective units of shame (SUS) at the end of the intervention | through study completion, an average of 3 months
  Subjective units of shame (SUS), taken at four points during the intervention (scored 0 no shame to 100 full of shame)

SECONDARY OUTCOMES:
Body Image States Scale | through study completion, an average of 3 months
  It will be used to assess transient feelings about the body and physical appearance. A 6-item scale measures current body-image experiences at a particular point in time or in a specific context. Possible scores range from 6 to 54, and higher scores indicate more positive body image (better outcome).
Shame subscale of the State Shame and Guilt Scale | through study completion, an average of 3 months
  It will be used to test state shame. Possible scores are ranged from 5 to 25. Higher scores indicate worse state shame.

CONTACTS AND LOCATIONS:
Locations (1):
- Fidan Turk, Sheffield, United Kingdom